CLINICAL TRIAL: NCT07097961
Title: Paediatric Post-TB Home-based Pulmonary Rehabilitation Feasibility Study
Brief Title: Paediatric Post-TB Pulmonary Rehab Study
Acronym: PPT Rehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: MU-JHU CARE (Other)
Responsible Party: Principal Investigator, Greta L. Becker, Resident Physician, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202503518; MHREC 2025-282 (Other: Mulago Hospital Research and Ethics Committee (MHREC)); HS622ES (Other: Uganda National Council for Science and Technology (UNCST))
Record Dates: First submitted 2025-07-13; First posted 2025-08-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Tuberculosis in Children; Chronic Lung Disease; Post Tuberculosis
Keywords: Post-TB lung disease; Uganda; Pulmonary rehabilitation; pediatric tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-Based Pulmonary Rehabilitation Program (Experimental)
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — The intervention includes twice-weekly walking and wall sit exercises, guided by a physiotherapy assessment. Participants use a pedometer, receive written instructions, and are monitored weekly by phone or home visit. Caregivers supervise the exercises and sessions are logged in a participant workbook.

SUMMARY:
The goal of this clinical trial is to learn if a home-based pulmonary rehabilitation program is feasible and acceptable for children ages 6-15 who have recently completed treatment for pulmonary tuberculosis. The main questions it aims to answer are:

Can children and caregivers follow a 6-week rehabilitation program?

Is the program acceptable and feasible for children and caregivers?

Researchers will also explore preliminary changes in walking distance and quality of life.

Participants will:

Attend a clinic visit for baseline testing, including a 6-minute walk test (6MWT) and the St. George's Respiratory Questionnaire (SGRQ)

Receive exercise instructions and a pedometer

Complete home-based walking and wall sit exercises twice per week for 6 weeks

Receive weekly follow-up from study staff (by phone or home visit)

Return to clinic at 6 weeks for follow-up testing

DETAILED DESCRIPTION:
An estimated 1.3 million children worldwide develop active tuberculosis (TB) annually, with pulmonary TB being the most common form. Even after successful treatment, children may experience persistent respiratory symptoms and long-term structural and functional lung damage, referred to as post-TB lung disease (PTLD). In Uganda, a high-burden TB and HIV country, the burden of PTLD in children is increasingly recognized, yet evidence-based management strategies are lacking.

PTLD can lead to significant impairments in lung function, exercise capacity, and quality of life. In a recent cross-sectional study conducted by the investigators, Ugandan children aged 6-16 years who had completed TB treatment were more likely to have abnormal lung function, radiographic abnormalities (e.g., fibrosis, pleural thickening), and reduced quality of life compared to household controls.

Pulmonary rehabilitation, a structured program of aerobic and strength exercises, has been shown to improve outcomes in adults with chronic lung disease, including PTLD, but has not been adapted or evaluated in children. This is particularly true in low-resource settings where facility-based programs are often inaccessible.

This single-arm feasibility study will assess the delivery of a 6-week home-based pulmonary rehabilitation program among children aged 6-17 years with previously diagnosed PTLD in Uganda. Participants will be recruited from an existing observational cohort or referred by clinicians based on prior TB history and persistent respiratory impairment. The program includes twice-weekly walking and strength exercises supervised by caregivers, guided by physiotherapy assessment. Weekly monitoring will be conducted through phone calls or home visits, and participants will track their activity using a pedometer and an exercise workbook.

The primary focus is to evaluate whether this intervention can be feasibly implemented in a pediatric population in a low-resource context and to inform the design of a future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-17 years
* Previously diagnosed with post-TB lung disease,
* Willing to remain in the study catchment area during the study period
* Able to participate in mild-to-moderate physical activity (late inclusion criterion)

Exclusion Criteria:

* Currently participating in another rehabilitation program
* Residence outside the Kampala metropolitan area
* Active respiratory infection (late exclusion criterion)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Adherence rate | 6 weeks
  Proportion of prescribed home-based exercise sessions (walking and strength) completed over the 6-week intervention period, as recorded in participant logbooks and verified during weekly follow-up.
Acceptability | 6 weeks
  Acceptability of the home-based pulmonary rehabilitation program as assessed by structured caregiver and participant feedback collected at the end of the 6-week intervention.

SECONDARY OUTCOMES:
Change in St. George's Respiratory Questionnaire (SGRQ) score | 6 weeks
  The absolute difference in SGRQ total score and sub-scores from baseline (enrollment visit) to the 6-week follow-up following pulmonary rehabilitation. The SGRQ is a validated tool used to assess health-specific quality of life.
Change in Six-Minute Walk Distance (6MWT) | 6 weeks
  The absolute difference in meters walked during the standardized 6MWT from baseline (enrollment visit) to the 6-week follow-up following pulmonary rehabilitation. The 6MWT is a validated test used to measure exercise capacity.
Change in Body mass index (BMI) | 6 weeks
  The difference in BMI-for-age Z-score, a standardized measure of body mass index adjusted for age and sex, from baseline to the 6-week follow-up. BMI is calculated as weight in kilograms divided by height in meters squared (kg/m²). Z-scores are computed using WHO child growth standards.

OTHER OUTCOMES:
Retention | 6 weeks
  The proportion of enrolled participants who complete the 6-week intervention and attend the follow-up visit. This measure provides information on the feasibility of participant follow-up.
Adverse events during intervention period | 6 weeks
  Number and type of adverse events (e.g., injury, worsening respiratory symptoms) reported during the 6-week rehabilitation program.
Change in walking session distance/steps across the 6-week intervention | 6 weeks
  Change in the distance walked during prescribed home-based walking sessions from the beginning to the end of the 6-week rehabilitation program, as recorded in participant logbooks. This outcome will explore trends in functional improvement during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Greta L Becker, MD, Principal Investigator — University of Iowa; Eric Wobudeya, MBChB, MMED, MSc, Principal Investigator — MU-JHU Care Ltd/MU-JHU Research Collaboration
Locations (1):
- MU-JHU Care Ltd/MU-JHU Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plan has not been finalized. The study team will consider sharing de-identified participant data upon request.

REFERENCES:
- [Background] Migliori GB, Marx FM, Ambrosino N, Zampogna E, Schaaf HS, van der Zalm MM, Allwood B, Byrne AL, Mortimer K, Wallis RS, Fox GJ, Leung CC, Chakaya JM, Seaworth B, Rachow A, Marais BJ, Furin J, Akkerman OW, Al Yaquobi F, Amaral AFS, Borisov S, Caminero JA, Carvalho ACC, Chesov D, Codecasa LR, Teixeira RC, Dalcolmo MP, Datta S, Dinh-Xuan AT, Duarte R, Evans CA, Garcia-Garcia JM, Gunther G, Hoddinott G, Huddart S, Ivanova O, Laniado-Laborin R, Manga S, Manika K, Mariandyshev A, Mello FCQ, Mpagama SG, Munoz-Torrico M, Nahid P, Ong CWM, Palmero DJ, Piubello A, Pontali E, Silva DR, Singla R, Spanevello A, Tiberi S, Udwadia ZF, Vitacca M, Centis R, D Ambrosio L, Sotgiu G, Lange C, Visca D. Clinical standards for the assessment, management and rehabilitation of post-TB lung disease. Int J Tuberc Lung Dis. 2021 Oct 1;25(10):797-813. doi: 10.5588/ijtld.21.0425. PMID 34615577
- [Background] Becker GL, Kisembo H, Sato Y, Wendt LH, Aanyu-Tukamuhebwa H, Nantanda R, Jackson JB, Blount RJ, Wobudeya E. Post-TB lung function, quality of life, and radiographic findings in children. IJTLD Open. 2025 Jul 9;2(7):427-433. doi: 10.5588/ijtldopen.24.0675. eCollection 2025 Jul. PMID 40657266
- See also: Makerere University-Johns Hopkins University Research Collaboration — https://www.mujhu.org/
- See also: University of Iowa Department of Internal Medicine Research Programs — https://medicine.uiowa.edu/internalmedicine/research